CLINICAL TRIAL: NCT05721768
Title: Altered Respiratory Compliance Under Invasive Mechanical Ventilation in SARS-CoV-2 & Development of Respiratory Sequels
Acronym: COMPLI-QUO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Simon VALENTIN, Principal investigator, University Hospital Practitioner, Pulmonology Department, Central Hospital, Nancy, France
Other Study IDs: 2022PI195
Record Dates: First submitted 2023-02-01; First posted 2023-02-10 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: ARDS Due to Disease Caused by SARS Co-V-2; Respiratory Compliance; Sequels of COVID

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal is to study the association between the value of the compliance of the respiratory system at the first day of the initiation of invasive mechanical ventilation and the presence of respiratory sequelae at a distance from the COVID-19 infection with the hypothesis that patients who have presented an alteration of the compliance of the respiratory system are at greater risk of developing respiratory sequelae.

Studying the altered compliance of the respiratory system in ARDS secondary to COVID-19 and its relationship to the development of respiratory sequelae would help us to improve the management of patients with COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized in intensive care medicine between 01/03/2030 and 01/09/2022 (with invasive mechanical ventilation for at least 48 hours for a SARS-CoV-2 infection documented by RT-PCR) who were followed in pulmonary outpatient medicine at least 3 months after their hospitalization in intensive care medicine and before 01/12/2022 and who had respiratory sequelae during this period.
* Hospitalized in intensive care medicine between 01/03/2020 and 01/12/2021 (with invasive mechanical ventilation for at least 48 hours for SARS-CoV-2 infection documented by RT-PCR) who were followed up in pulmonary outpatient medicine but did not have respiratory sequelae between 01/06/2020 and 01/12/2022.

Exclusion Criteria:

* Documented underlying respiratory pathology.
* Pneumothorax within the first 10 days.
* Patient requiring extracorporeal circulatory support.
* Refusal to participate
* Persons referred to in articles L. 1121-5, L. 1121-7 and L1121-8 of the public health code: Pregnant woman, parturient or breastfeeding mother / Minor (not emancipated) / Adult subject to a legal protection measure (guardianship, curatorship, safeguard of justice) / Adult unable to express his consent
* Persons deprived of liberty by a judicial or administrative decision, persons under psychiatric care under articles L. 3212-1 and L. 3213-1.
* Respiratory system compliance data not available on the computer software

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients followed in the Outpatient Medicine Unit of the Respiratory Department of the Nancy University Hospital in the framework of the post COVID-19 follow-up, previously hospitalized in intensive care medicine and intensive care unit.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-02-24 (Actual); Primary Completion 2023-03-15 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Presence of respiratory sequelae | 1 year
  Presence of respiratory sequelae (FVC <80% or DLCO <70% or radiologic sequelae attributable to SARS-CoV-2) at M3 or M6 or M12

CONTACTS AND LOCATIONS:
Locations (1):
- Valentin Simon, Nancy, France

IPD SHARING:
Plan to Share IPD: No